CLINICAL TRIAL: NCT06325774
Title: Safety and Efficacy Study of Hypofractionated Radiotherapy for Localized Prostate Cancer: a Single-arm Clinical Trial
Brief Title: Radical Hypofractionated Radiotherapy for Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Changhai HHospital
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Localized Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Radiotherapy (Experimental): Hypofractionated Radiotherapy over 3 weeks.
  Interventions: Radiation: Hypofractionated radiation therapy

INTERVENTIONS:
Radiation: Hypofractionated radiation therapy — 54 Gy in 15 daily fractions of 3.6 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.

SUMMARY:
The aim of this trial is to study the safety outcomes of hypofractionated radiotherapy in treating patients with localized prostate cancer.

Hypofractionated radiotherapy delivers higher doses of radiotherapy in a shorter time period, may enabling the killing of more tumor cells with fewer side effects.

Accumulating evidence has proven the safety and feasibility of hypofractionated radiotherapy for localized prostate cancer.But for localized prostate cancer,the optimal dose per fraction of hypofractionated radiotherapy is still on its way.

DETAILED DESCRIPTION:
The present study will be conducted as a prospective, open-label, single-arm clinical trial.

The patients will receive hypofractionated radiation(54 Gy in 15 daily fractions of 3.6 Gy ). After completion of study treatment, patients were followed up once a month for the first 3 months and once every 3 months after 3 months for a total of 5 years.

The primary endpoints of the study are the toxicities about gastrointestinal (GI),genitourinary (GU) symptoms and erectile dysfunction.The secondary endpoints include progression-free survival (bPFS), local progression-free-survival(LPFS) ,distant metastasis free survival(DMFS) ,overall survival (OS)and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old;
* European Cooperative Oncology Group score(ECOG):≤ 2;
* Patients with pathologically diagnosed prostate cancer;
* Clinical stage was cTanyN0M0 any Gleason / ISUP group;
* Expected survival time >5 years;
* The patient has no contraindications to radiotherapy and is suitable and willing to undergo radiotherapy;
* Patients who voluntarily accept the experimental study protocol after being informed about the existing treatment options;

Exclusion Criteria:

* Patients who have received any other early treatment for prostate cancer, including radiotherapy, chemotherapy, focal therapy, etc;
* a previous history of pelvic and abdominal radiotherapy;
* Prior hormonal therapy (castration or antiandrogen);
* Patients with other malignancies and acute or chronic infections such as human immunodeficiency virus (HIV) (+), hepatitis C virus (HCV) (+) and/or positive syphilis;
* Patients that the investigator considers unsuitable to participate in the clinical trial; patients with other serious systemic diseases, evaluation and compliance of the trial, including severe respiratory, circulatory, neurological, mental, digestive, endocrine, immune, urinary, and other systemic diseases;
* Patients with contraindications related to radiotherapy;
* Participate in other clinical trials that are mutually exclusive with the study intervention within 4 weeks prior to the start of the study;
* Patients unable to provide written informed consent or demonstrate poor treatment compliance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiotherapy-related gastrointestinal and urogenital tract adverse events | 5 years
  RTOG / EORTC scale, Common Terminology Criteria for Adverse Events (CTCAE) 5.0, erectile dysfunction.

SECONDARY OUTCOMES:
biochemical progression-free survival (bPFS) | 5 years
  The definition of biochemical failure is a PSA measurement ≥ PSA nadir + 2 ng/mL where nadir is the lowest post-RT PSA value.Time to biochemical failure is defined as time from randomization to the date of first biochemical failure, last known follow-up (censored), or death without biochemical failure (competing risk).
local progression-free-survival(LPFS) | 5 years
  Response evaluation criteria in solid tumor（RECIST）1.1:To determine the outcome of treatment for solid tumors,The efficacy according the diameter of the lesion could be divided into complete response（CR），partial response（PR）,stable disease（SD）and progressive disease（PD）.
distant metastasis free survival(DMFS) | 5 years
  Distant metastasis (failure) is defined as radiographic evidence of hematogenous spread evaluated by bone scan, CT, or MRI. Time to distant metastasis is defined as time from randomization to the date of first distant metastasis, last known follow-up (censored), or death without local recurrence (competing risk).
Overall survival (OS) | 5 years
  Overall survival time is defined as time from registration/randomization to the date of death (failure) from any cause or last known follow-up (censored).
Quality of life (QoL) | 5 years
  Expanded Prostate Cancer Index (EPIC-26)：The EPIC is a prostate cancer health-related quality of life (HRQOL) self-administered instrument measuring patient-reported urinary, bowel, sexual, and hormonal symptoms related to prostate cancer treatments. Response options for each item form a Likert scale with scores transformed linearly to a 0-100 scale. Domain scores are also on a 0-100 scale with higher scores representing better HRQOL.
Physical Activity Rank Scale-3 (ARS-3) | 5 years
  To assess the physical activity rank.The scale was compiled by Japanese psychologist KIMIO HASHIMOTO and introduced and revised by Liang Deqing from Wuhan Physical Education University. There are only 3 items in this scale, which adopts 5 grades from 1 to 5, and examines the level of physical activity from 3 aspects: intensity, time and frequency of participating in physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists and specialists in surgerywho are interested in examining the efficacy and toxicity of localized prostate cancer treated with radical hypofractionated radiotherapy. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.

REFERENCES:
- [Derived] Liang Y, Zhang W, Zhao X, Zhang H. Hypofractionated radiotherapy for localized prostate cancer: the protocol for a prospective clinical trial. Future Oncol. 2025 May;21(12):1483-1488. doi: 10.1080/14796694.2025.2489340. Epub 2025 Apr 21. PMID 40257456